CLINICAL TRIAL: NCT02786550
Title: Botulinum Toxin to Improve Lower Blepharoplasty Scar
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 104-8788A3
Record Dates: First submitted 2016-05-26; First posted 2016-06-01 (Estimated); Last update posted 2016-06-23 (Estimated); Status verified 2016-05

CONDITIONS: Other Degenerative Disorders of Eyelid and Periocular Area
Keywords: Lower blepharoplasty, Botulinum toxin, Scar
MeSH Terms: conditions — Cicatrix | interventions — Botulinum Toxins; Botulinum Toxins, Type A; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Botulinum Toxin (Experimental): Immediately after lower blepharoplasty surgery 3 injections of 2.5U of botulinum toxin over lateral part of orbicularis oculi muscle.
  Intervention: Botulinum toxin injection
  Interventions: Drug: Botulinum Toxin
- Normal saline (Placebo Comparator): Immediately after lower blepharoplasty surgery 3 injections of same amount of normal saline over lateral part of orbicularis oculi muscle.
  Intervention: Normal saline injection
  Interventions: Other: Normal Saline

INTERVENTIONS:
Drug: Botulinum Toxin — A total of 7.5U per side of botulinum toxin will be injected to the lateral part of obicularis oculis muscle (3 injections of 2.5 U).
  Other Names: Botulinum Toxin Type A; Botox
  Arms: Botulinum Toxin
Other: Normal Saline — The same amount (3 cc) of Normal saline will be injected to the lateral part of obicularis oculis muscle
  Other Names: Na Cl 0.9%
  Arms: Normal saline

SUMMARY:
The combination of Botulinum toxin for crow feet (lateral part of orbicularis oculi muscle) and lower blaphaloplasty might have reduces the tension on the end of lower blaphaloplasty incision whereas the scar is more visible on patient.

The main aim of this trial is to investigate whether the injection of Botulinum toxin into the bilateral orbicularis oculi muscles could improve the appearance of the scar after lower blepharoplasty.

DETAILED DESCRIPTION:
The main aim of this double blind randomized trial is to examine whether immediate post-operative injection of botulinum toxin into lateral part of bilateral orbicularis oculis muscles (the injection technique of crow feet) can improve scar formation for lower blepharoplasty patients.

This is a double blind randomized controlled trial primarily designed to compare the scarring after secondary cleft lip repair with immediate post-operative botulinum toxin injection into the into bilateral lateral orbicularis oculi muscles in patients with lower blepharoplasty. There will be 2 main groups in this study:-

1. Study group (Group I): Immediately after lower blepharoplasty surgery 3 injections of 2.5U of botulinum toxin over lateral part of orbicularis oculi muscle.
2. Control group (Group II): There will be the same amount of normal saline injection after lower blepharoplasty.

Follow-up Assessments Vancouver scar scale measures pigmentation, vascularity, pliability and scar height on the postoperative 6 month Follow Up.

Visual analogue scale They were asked to score the scars on the photographs using a standard visual analogue scale graded from 0 (worst possible scar) to 10 (best possible scar).

Photographic measurement:

A ruler will be placed just below the surgical scar. Using Photoshop CS5, the scar width can be measured.

Chi-square will be used to analyze the demographic data ( i.e. Gender) The Independent T-Student test will be used to analyze the statistical significance between the two groups.

The dosage of Botox that the investigators use for crowfeet is very tiny. And this is a common clinic practice. Systemic insult is unlikely to happen. If an allergic reaction occurred it will be treated according to the severity of allergy and Diphenhydramin PO or IV form or systemic corticosteroid will be given.

ELIGIBILITY:
Inclusion Criteria:

1. Adult ≥ 45 years old.
2. Lower eyelid Rhytidosis and dermatochalasis.
3. Lower eyelid steatoblepharon and pronounced nasojugal groove
4. Written informed consent given by patient.

Exclusion Criteria:

1. Less than 45 years old
2. Without written informed consent.
3. Combined other craniofacial anomalies

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2016-06; Primary Completion 2018-06 (Estimated); Study Completion 2018-06 (Estimated)

PRIMARY OUTCOMES:
Visual analogue scale | 6 months after surgery
  to score the scars on the photographs using a standard visual analogue scale graded from 0 (worst possible scar) to 10 (best possible scar).

SECONDARY OUTCOMES:
Vancouver scar scale | 6 months after surgery
  Use vancouver scar scale to access the scar of blepharoplasty
Photographic measurement | 6 months after surgery
  A ruler will be placed just below the surgical scar. Using Photoshop CS5, the scar width can be measured

CONTACTS AND LOCATIONS:
Overall Officials: Henry Yau-Li Huang, M.D., Principal Investigator — Department of Dermatology, Chang Gung Memorial Hospital
Locations (1):
- Chun-Chin Chang, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Chang CS, Wallace CG, Hsiao YC, Chang CJ, Chen PK. Botulinum toxin to improve results in cleft lip repair: a double-blinded, randomized, vehicle-controlled clinical trial. PLoS One. 2014 Dec 26;9(12):e115690. doi: 10.1371/journal.pone.0115690. eCollection 2014. PMID 25541942
- [Background] Chang CS, Wallace CG, Hsiao YC, Chang CJ, Chen PK. Botulinum toxin to improve results in cleft lip repair. Plast Reconstr Surg. 2014 Sep;134(3):511-516. doi: 10.1097/PRS.0000000000000416. PMID 25158709
- [Background] Zhang DZ, Liu XY, Xiao WL, Xu YX. Botulinum Toxin Type A and the Prevention of Hypertrophic Scars on the Maxillofacial Area and Neck: A Meta-Analysis of Randomized Controlled Trials. PLoS One. 2016 Mar 17;11(3):e0151627. doi: 10.1371/journal.pone.0151627. eCollection 2016. PMID 26985661
- [Background] Lee SJ, Jeong SY, No YA, Park KY, Kim BJ. Combined Treatment with Botulinum Toxin and 595-nm Pulsed Dye Laser for Traumatic Scarring. Ann Dermatol. 2015 Dec;27(6):756-8. doi: 10.5021/ad.2015.27.6.756. Epub 2015 Dec 7. PMID 26719648
- [Background] Prodromidou A, Frountzas M, Vlachos DE, Vlachos GD, Bakoyiannis I, Perrea D, Pergialiotis V. Botulinum toxin for the prevention and healing of wound scars: A systematic review of the literature. Plast Surg (Oakv). 2015 Winter;23(4):260-4. doi: 10.4172/plastic-surgery.1000934. PMID 26665143
- [Background] Zelken J, Yang SY, Chang CS, Chang CJ, Yang JY, Chuang SS, Chen HC, Hsiao YC. Donor Site Aesthetic Enhancement With Preoperative Botulinum Toxin in Forehead Flap Nasal Reconstruction. Ann Plast Surg. 2016 Nov;77(5):535-538. doi: 10.1097/SAP.0000000000000625. PMID 26418784